CLINICAL TRIAL: NCT02862769
Title: The Role of Intra-operative Lidocaine Infusion in Preventing Chronic Post Surgical Pain After Video Assisted Thoracoscopic Surgery
Brief Title: Intra-operative Lidocaine Infusion in Preventing CPSP Post VATs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Qutaiba Tawfic, MD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSREB 107989
Record Dates: First submitted 2016-07-28; First posted 2016-08-11 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Chronic Pain; Acute Pain; Neuralgia
MeSH Terms: conditions — Chronic Pain; Acute Pain; Neuralgia | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine infusion (Experimental): first group (lidocaine group) will include those who receive a intraoperative lidocaine infusion (Induction bolus dose of 1.5 mg/kg body weight followed by a continous lidocaine infusion
  Interventions: Drug: Lidocaine
- Saline Infusion (Placebo Comparator): The second group will include those who receive a intraoperative placebo i(Induction bolus dose of 1.5 mg/kg body weight of lidocaine followed by a continous saline infusion at the same rate as the lidocaine infusion.
  Interventions: Drug: Lidocaine; Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — . Perioperatively, when lidocaine is administered as a continuous infusion at clinically relevant doses (1-2 mg/kg/hr) results in plasma concentration below 5µg.mL-1. At this plasma level, it is adequate to attenuate sympathetic responses , decrease pain and demonstrate a significant opioid sparing effect.
Drug: Saline — The second group will include those who receive a intraoperative placebo infusion(saline infusion) (Induction bolus dose of 1.5 mg/kg body weight followed by a continous saline infusion 1.5 mg/kg/hr.
  Arms: Saline Infusion

SUMMARY:
The aim of this study is to evaluate the impact of intravenous lidocaine on acute and chronic post surgical pain on patients undergoing video assisted thoracoscopic surgery(VATS). The investigators believe that systemic administration of lidocaine during the perioperative period would be effective in preventing chronic pain post VATS. In addition to chronic pain the investigators believe it will reduce acute postoperative pain as well as each patients total opioid requirement.The investigators believe that this will have a significant impact on the care of patients presenting for VATS.

DETAILED DESCRIPTION:
It is not surprising that complications related to surgical procedures occur. Chronic Post Surgical Pain (CPSP) is considered one of the more common surgical complications, despite all the advances in understanding acute pain and the development of new modalities for pain management 1. Chronic Post Surgical Pain was defined by Macrae and Davies 7 as a persistent pain, which existed for a minimum of two months following a surgical procedure. The condition of pre-existence of pain, and causes for the pain other than surgery should be excluded. Thoracic surgeries including thoracotomy and video-assisted thoracoscopic surgery (VATS) are some of the highest risk procedures that often lead to CPSP. The prevalence of chronic pain after VATS is close to that after thoracotomy (25-47 %), half of them having neuropathic pain A, B. Because of the fact that chronic pain is a major physical and mental health care problem affecting the patient and the community in general, it has become essential for physicians to prevent the development of chronic pain 8.

While multimodal analgesia has largely replaced pain mono-therapy with opioids, they remain the most commonly used medications to treat post operative pain. Lidocaine is an amide local anesthetic which when used intravenously demonstrates significant analgesic, anti-hyperalgesic and anti-inflammatory properties . It also reduces the sensitivity and activity of spinal cord neurons, decreases N-methyl-D-aspartate (NMDA) receptors mediated post-synaptic depolarization. The analgesic effects of systemic lidocaine were first tested in chronic neuropathic pain when the results support the usage of these drugs. Perioperatively, when lidocaine is administered as a continuous infusion at clinically relevant doses (1-2 mg/kg/hr) results in plasma concentration below 5µg.mL-1. At this plasma level, it is adequate to attenuate sympathetic responses , decrease pain and demonstrate a significant opioid sparing effect. Perioperative lidocaine administration was associated with a decreased incidence of CPSP when it is associated with neuropathic pain . It reduced CPSP in mastectomy by 40-50% after 3 and 6 months follow-up. To the best of our knowledge there is no study that has addressed the usage of lidocaine in VATS or thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* VATs for lobectomy
* Understanding of English (reading, writing and speaking)
* Written consent for being involved in this study
* Exclusion Criteria:
* Chronic pain including fibromyalgia
* Patients using opioids (more than 80 mg equivalent of oral morphine/day for >60 days)
* Major depression
* Received or going to receive chemotherapy or radiotherapy.
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Chronic Pain post VATs | 3 months
  Using the Brief Pain Inventory Scale
Chronic Pain post VATs | 6 months
  Using the Brief Pain Inventory Scale

SECONDARY OUTCOMES:
Opioid requirement | 48 hours
  Calculating Opioid dose(1hr, 6hr, 24 hrs and 48 hrs)
Pain Score for Acute Post Operative Pain | 48 hours post-op
  Using Numerical Pain Scale
Mean Pain Scores | 3 and 6 months
Pain interference | 3 and 6 months
  Using the Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Qutaiba Tawfic Hamodi, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruce J, Quinlan J. Chronic Post Surgical Pain. Rev Pain. 2011 Sep;5(3):23-9. doi: 10.1177/204946371100500306. PMID 26526062
- [Result] Steegers MA, Snik DM, Verhagen AF, van der Drift MA, Wilder-Smith OH. Only half of the chronic pain after thoracic surgery shows a neuropathic component. J Pain. 2008 Oct;9(10):955-61. doi: 10.1016/j.jpain.2008.05.009. Epub 2008 Jul 16. PMID 18632308
- [Result] Peng Z, Li H, Zhang C, Qian X, Feng Z, Zhu S. A retrospective study of chronic post-surgical pain following thoracic surgery: prevalence, risk factors, incidence of neuropathic component, and impact on qualify of life. PLoS One. 2014 Feb 28;9(2):e90014. doi: 10.1371/journal.pone.0090014. eCollection 2014. PMID 24587187
- [Result] Usichenko TI, Rottenbacher I, Kohlmann T, Julich A, Lange J, Mustea A, Engel G, Wendt M. Implementation of the quality management system improves postoperative pain treatment: a prospective pre-/post-interventional questionnaire study. Br J Anaesth. 2013 Jan;110(1):87-95. doi: 10.1093/bja/aes352. Epub 2012 Oct 9. PMID 23048069